CLINICAL TRIAL: NCT04184128
Title: Prevalence of Detrusor Underactivity and Bladder Outlet Obstruction in Women With Cystocele and Changes of Voiding Function After Cystocele
Brief Title: Detrusor Underactivity and Bladder Outlet Obstruction in Women With Cystocele
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907008RINC
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-07

CONDITIONS: Cystocele
Keywords: Bladder outlet obstruction; Detrusor underactivity; Cystocele
MeSH Terms: conditions — Cystocele; Urinary Bladder Neck Obstruction; Urinary Bladder, Underactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Detrusor underactivity: The DU was defined when the PdetQmax was less than 20 cmH2O, the Qmax was less than 15 mL/s, and the bladder voiding efficiency (BVE) was less than 90 %. BVE = voided volume / (voided volume+ PVR) x 100%.
  Interventions: Diagnostic Test: Urodynamic study
- Bladder outlet obstruction: The BOO was defined when the PdetQmax was not less than 40 cmH2O, and the Qmax was less than 12 mL/s.
  Interventions: Diagnostic Test: Urodynamic study
- Non-DU/BOO group: Those women without DU or BOO were allocated to the non-DU/BOO group.
  Interventions: Diagnostic Test: Urodynamic study

INTERVENTIONS:
Diagnostic Test: Urodynamic study — The urodynamic assessment included uroflowmetry, filling cystometry with 35°C distilled water at a rate of 60 mL/sec, a pressure flow study, and a stress urethral pressure profile with patient in sitting position [14]. A 20-minute pad test for each woman was also performed [15, 16]. Multichannel urodynamic equipment (Life-Tech, Houston, TX, USA) with computer analysis and Urovision (Urolab Janus System V, Houston) was used. All terminology conformed to the standards recommended by the ICS [3]. All procedures were performed by an experienced technician, and the data were interpreted by a single observer to avoid interobserver variability.
  Other Names: Pad test

SUMMARY:
Women with cystocele may be associated with detrusor underactivity (DU) or bladder outlet obstruction (BOO). However, the impact of cystocele repair on the rates of DU and BOO remained obscure. Thus, the aim of this study was to elucidate the prevalence of DU and BOO in each age group and elucidate the impact of cystocele repair on the rates of DU and BOO.

DETAILED DESCRIPTION:
Between November 2010 and September 2018, all women with ≥ POP-Q stage II cystocele who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed. Those women who have no complete data of maximum flow rate (Qmax), voided volume, post-void residual volume (PVR) and detrusor pressure at a maximum flow rate (PdetQmax) were excluded from this study. The DU was defined when the PdetQmax was less than 20 cmH2O, the Qmax was less than 15 mL/s, and the bladder voiding efficiency (BVE) was less than 90 %. The BOO was defined when the PdetQmax was not less than 40 cmH2O, and the Qmax was less than 12 mL/s. BVE = voided volume / (voided volume+ PVR) x 100%. Those women without DU or BOO were allocated to the non-DU/BOO group.

STATA software was used for statistical analysis. Wilcoxon signed-rank test or McNemar's test was used for statistical analysis as appropriate. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ≥ POP-Q stage II cystocele
* Female

Exclusion Criteria:

* Those women who have no complete data of maximum flow rate (Qmax), voided volume, post void residual volume (PVR) and detrusor pressure at maximum flow rate (PdetQmax) were excluded from this study.

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All medical records of women with ≥ POP-Q stage II cystocele who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
DU or BOO | Between November 2010 and September 2018
  The DU was defined when the PdetQmax was less than 20 cmH2O, the Qmax was less than 15 mL/s, and the bladder voiding efficiency (BVE) was less than 90 % [1]. The BOO was defined when the PdetQmax was not less than 40 cmH2O, and the Qmax was less than 12 mL/s [1]. BVE = voided volume / (voided volume+ PVR) x 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Result] Lamblin G, Delorme E, Cosson M, Rubod C. Cystocele and functional anatomy of the pelvic floor: review and update of the various theories. Int Urogynecol J. 2016 Sep;27(9):1297-305. doi: 10.1007/s00192-015-2832-4. Epub 2015 Sep 4. PMID 26337427
- [Result] Frigerio M, Manodoro S, Cola A, Palmieri S, Spelzini F, Milani R. Detrusor underactivity in pelvic organ prolapse. Int Urogynecol J. 2018 Aug;29(8):1111-1116. doi: 10.1007/s00192-017-3532-z. Epub 2017 Dec 21. PMID 29270721
- [Result] Hsiao SM, Lin HH, Kuo HC. Videourodynamic Studies of Women with Voiding Dysfunction. Sci Rep. 2017 Jul 28;7(1):6845. doi: 10.1038/s41598-017-07163-2. PMID 28754926
- [Result] Huang WC, Yang SH, Yang JM. Clinical Importance and Surgical Outcomes of Green Type III Cystocele in Women With Anterior Vaginal Prolapse. J Ultrasound Med. 2015 Dec;34(12):2279-85. doi: 10.7863/ultra.14.11066. Epub 2015 Nov 16. PMID 26573101
- [Result] Salinas Casado J, Adot Zurbano JM, Dambros M, Virseda Chamorro M, Ramirez Fernandez JC, Moreno Sierra J, Marcos Diaz J, Silmi Moyano A. [Factors for voiding dysfunction and cystocele]. Arch Esp Urol. 2005 May;58(4):316-23. doi: 10.4321/s0004-06142005000400006. Spanish. PMID 15989095